CLINICAL TRIAL: NCT01535092
Title: A Randomized, Double-Blind, Placebo Controlled Study to Investigate the Efficacy and Safety of Legalon SIL for the Treatment of HCV Recurrence of the Graft in Orthotopic Liver Transplant Patients
Brief Title: Legalon SIL for the Treatment of HCV Recurrence in Liver Transplanted Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: when realized that the target 60% of patients with SVR was no more achievable
Sponsor: Rottapharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEG-SIL-LTX-03
Record Dates: First submitted 2012-02-07; First posted 2012-02-17 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: HCV Recurrence After Liver Transplantation
Keywords: HCV recurrence; HCV reinfection; Liver transplantation; Legalon SIL; silibinin; viral load
MeSH Terms: interventions — Silybin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- silibinin (Experimental): Silibinin 20mg/Kg/day (Legalon SIL) by intravenous infusion for 14-21 days before OLT and for 7 days after OLT
  Interventions: Drug: Silibinin
- Placebo (Placebo Comparator): Placebo (NaCl 0.9% - saline) administered daily by intravenous infusion for 14-21 days before OLT and 7 days after OLT
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Silibinin — 20mg/Kg daily by intravenous infusion, for 14-21 days pre-OLT and for 7 days post-OLT
  Other Names: Legalon SIL
  Arms: silibinin
Drug: Placebo — Saline, daily infused for 14-21 days pre-OLT and for 7 days post-OLT
  Arms: Placebo

SUMMARY:
Orthotopic liver transplantation (OLT) is the treatment of choice for patients with Hepatitis C Virus (HCV) infection and end-stage liver disease or hepatocellular carcinoma; infection of the graft and hepatitis C recurrence is universal after OLT and recurrent HCV hepatitis often follows an accelerated course after OLT, with rapid histological recurrence and cirrhosis. These very poor outcome significantly affect graft and patient survival and reduces the benefit of transplantation for this indication. Therapeutic strategies are not available; high viral load, high prevalence of genotype 1b and need of dose reduction of interferon and ribavirin because of the side effects or intolerance, together with the interference of immunosuppressive drugs, resulted in the vast majority of the patients in failure in obtaining viral eradication.

Recently, Silibinin, has been studied and reported to be capable to act as potent antiviral agent in patients with HCV; it has been used successfully in a protocol of a 14 day intravenous infusion in previous non-responders to peginterferon/ribavirin therapy. In view of his postulated profile of safety, it seems an ideal drug to be used in the setting of HCV recurrent patients after liver transplant.

Aim of this prospective, randomized, double-blind, placebo-controlled, parallel group study is to determine the therapeutic effect of Legalon SIL in the prevention of HCV reinfection in chronically infected hepatitis C patients after OLT.

Awaiting orthotopic liver transplantation patients affected by HCV will be randomised 3:1 to receive, in addition to their current therapy, silibinin 20mg/kg/day (Legalon SIL) or placebo infused over 2 hours from 14 to 21 consecutive days; in addition, patients will receive treatment with silibinin 20mg/kg/day (Legalon SIL), infused over 2 hours, for 7 days after transplant.

The Primary Efficacy endpoint is to achieve sustained virological response (SVR) while Secondary Efficacy endpoints are to evaluate the virologic response, the percentage of patients who has a decreased of at least 2 log10 the levels of HCV-RNA and the safety of Legalon SIL in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must provide signed and dated informed consent before undergoing any trial related procedure.
2. Patient between 18 and 70 years of age.
3. Patient must have documented HCV infection. The HCV-RNA result obtained from the local laboratory at the screening visit must confirm HCV-RNA > 1000 IU/mL.
4. Patient must qualify for liver transplantation at the time of Screening according to Model for End stage Liver Disease (MELD) criteria
5. Patient must have a documented diagnosis of cirrhosis.
6. Patient weigh between 50 kg and 100 kg.
7. Patients must be able to communicate, participate and comply with the requirements of the entire study.
8. Female patients of child-bearing potential must agree on using a contraceptive method (oral contraceptive, intrauterine device, transdermal contraceptive patch) and must have a negative pregnancy urine test at screening.
9. HCV Genotype, chest X-ray, ultrasonography and ocular examination (for patients with history of diabetes or hypertension) must be performed within 6 months prior to Screening or between Screening and Day 1. 12-Lead ECG must be performed within 3 months prior to Screening.

Exclusion Criteria:

1. Patients known to be coinfected with the human immunodeficiency virus (HIV) or hepatitis B virus (HBsAg positive).
2. Active septic infections at time of screening.
3. Previous organ transplantation other than cornea and hair.
4. Use of systemic immunosuppressant or immunomodulating agents (including systemic corticosteroids) within 4 weeks of the screening visit or during the screening period.
5. Treatment for HCV with any investigational medication (prior use of silymarin is not exclusionary)
6. Treatment for HCV with any licensed therapies or prior maintenance therapy with any interferon alpha within 30 days of the randomization visit.
7. Participation in any other clinical trial within 30 days of randomization or intention to participate in another clinical trial during participation in this study.
8. Any known pre-existing medical condition that could interfere with the subject's participation in and completion of the study including but not limited to:

   * Chronic pulmonary disease (eg, clinical chronic obstructive pulmonary disease, interstitial lung disease, pulmonary fibrosis, sarcoidosis).
   * Current or history of any clinically significant cardiac abnormalities/dysfunction (eg, angina, congestive heart failure, myocardial infarction, pulmonary hypertension, complex congenital heart disease, cardiomyopathy, significant arrhythmia) including current uncontrolled hypertension, or history of use of antianginal agents for cardiac conditions.
   * Any other condition which, in the opinion of a physician-investigator, would make the patient unsuitable for enrollment or could interfere with the subject participating in and completing the study.
9. Subjects who are part of the site personnel directly involved with this study or those who are family members of the investigational study staff.
10. If female, pregnancy or breast-feeding.
11. Known hypersensitivity to Legalon® SIL.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Sustained virological response (SVR), defined as Virological Response (undetectable HCV-RNA) that lasts 6 months after the transplant | 6 months

SECONDARY OUTCOMES:
Virologic response (VR) defined as undetectable HCV RNA | after 14-21 days of pre-OLT and 7 days of post-OLT treatment; week 2, 3, 4, 8, 12, 24 after OLT
Percentage of patients who has a decreased of at least 2 log10 the levels of HCV-RNA | at week 4 after OLT
Number of patients with AE | after 14-21 days of pre-OLT and 7 days of post-OLT treatment; week 2, 3, 4, 8, 12, 24 after OLT
laboratory parameters | after 14-21 days of pre-OLT and 7 days of post-OLT treatment; week 2, 3, 4, 8, 12, 24 after OLT
blood levels of immunosuppressive drugs | week 1, 2, 3, 4, 8, 12, 24 after OLT
Vital signs | after 14-21 days of pre-OLT and 7 days of post-OLT treatment; week 2, 3, 4, 8, 12, 24 after OLT
ECG | after 14-21 days of pre-OLT and 7 days of post-OLT treatment; week 2, 3, 4, 8, 12, 24 after OLT

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Forns, Dr, Principal Investigator — Hospital Clinic i Barcelona